CLINICAL TRIAL: NCT05570331
Title: Clinical Evaluation of HPV Integration Triage for Detection of Cervical Precancer in HPV-positive Women：a Prospective Cohort Study
Brief Title: Clinical Evaluation of HPV Integration Triage for Detection of Cervical Precancer in HPV-positive Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ding Ma (Other)
Responsible Party: Sponsor-Investigator, Ding Ma, Chairman of Obstetrics & Gynecology department of Tongji hospital, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20220142
Record Dates: First submitted 2022-10-05; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: HPV Infection; Cervical Cancer
Keywords: Cervical cancer screening, HPV test, HPV integration
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical Exfoliated Cells sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HPV integration test — HPV-positive patients who are eligible for cervical cancer screening will be asked to collect Cervical Exfoliated Cells sample for the HPV integration screening test and for the HPV testing and TCT.

SUMMARY:
The American Society for Colposcopy and Cervical Pathology (ASCCP) recommended HPV testing or co-cytology testing as the standard primary approach for cervical cancer (CC) screening, which is highly sensitive for detection of cervical intraepithelial neoplasia grade 3 or worse. However, in clinical CC screening practice, the specificity and positive predictive value of the ASCCP-recommended strategy is relatively low, which leads to excessive colposcopy and common overtreatment, especially in China with a large number of cervical cancer cases. HPV integration in the host genome is a critical step in cervical carcinogenesis and is highly specific for detection of cervical cancer. Whether HPV integration analysis can play a role in the triage of cervical cancer screening has not yet been investigated.

DETAILED DESCRIPTION:
Based on the dilemma of the cervical cancer screening process, in the last five years, our team developed a novel cervical cancer triage strategy and conducted a large cohort study, which evaluated the clinical performance of HPV integration triage alone and in combination with HPV16/18 or HPV16 genotyping of HPV-positive women. We found that the specificity of HPV integration for greater than cervical intraepithelial neoplasia 3 was 94.5%, which was significantly higher than that of cytology (63.8%; P < 0.001) in our previous retrospective study.Here, we conducted a large prospective cohort study evaluating the clinical performance of HPV integration triage of HPV-positive women.

ELIGIBILITY:
Inclusion Criteria:

* Consenting women aged 20y-70y with HPV-positive results

Exclusion Criteria:

* Not providing informed consent
* previously confirmed CIN, cervical cancer, or other malignancies
* previous therapeutic procedure to cervix
* pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aged 20y-70y HPV-positive women
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of CIN2+ disease | 3 years
  CIN2+ diagnosed on biopsy obtained at colposcopy.
Risk of CIN3+ disease | 3 years
  CIN3+ diagnosed on biopsy obtained at colposcopy.

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD, PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided